CLINICAL TRIAL: NCT01868347
Title: The Obese Patient in the Urologic Robotic Surgery: the Role of a Preemptive Ventilator Strategy and Partitioning to Contrast Pneumoperitoneum and Trendelenburg Position
Brief Title: Obese Patient During RARP: the Role of a Preemptive Ventilator Strategy to Contrast Pneumoperitoneum and Trendelenburg Position
Acronym: OPERA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, PierPaolo Terragni, MD, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-20686
Record Dates: First submitted 2013-05-23; First posted 2013-06-04 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: Obese Patients With Prostate Cancer Disease
Keywords: obese patients; specific elastance; Trendelenburg Position; Pneumoperitoneum; robotic surgery; Prostatectomy
MeSH Terms: conditions — Pneumoperitoneum | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): PEEP after pneumoperitoneum and trendelenburg
  Interventions: Other: control
- Treatment (Experimental): preemptive PEEP before pneumoperitoneum and trendelenburg
  Interventions: Other: treatment

INTERVENTIONS:
Other: treatment — preemptive PEEP before pneumoperitoneum and trendelenburg
  Arms: Treatment
Other: control — PEEP after pneumoperitoneum and trendelenburg
  Arms: control

SUMMARY:
Analysis of the specific elastance during general anesthesia in patients treated with RARP (robotic assisted radical prostatectomy), to evaluate the efficacy of the preemptive strategy, involving recruitment maneuver and setting of 10 cmH2O PEEP before induction of pneumoperitoneum and trendelenburg position.

DETAILED DESCRIPTION:
RARP (robotic assisted radical prostatectomy) requires the induction of pneumoperitoneum and the trendelenburg position, causing increase in the intra-abdominal pressure and cephalic shift of the diaphragm, with consequent airway closure and collapse of the dependent regions of the lung.

Obese subjects present an increased risk of respiratory complications, caused not only by the surgical procedure itself, but also by the respiratory mechanics changes associated with the body mass. In obese patients we can observe higher values of lung and chest wall elastance, with reduction in ventilation-perfusion ratio.

The partitioning between lung and chest wall elastance can improve ventilatory setting and mechanics parameters of ventilation.

In every patient we will place, after anesthesia induction, a catheter to get esophageal and gastric pressure that represent pleural and abdominal pressure.

Ventilation will be conducted with a tidal volume of 8-10 ml/kg (IBW) and a respiratory rate adequate to maintain a physiological level of Pa CO2.

The preemptive strategy involves recruitment maneuver and setting of 10 cmH2O PEEP before induction of pneumoperitoneum and trendelenburg position in the treatment group, while the current procedure provides it afterwards (control group).

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 30
* Robotic-assisted laparoscopic prostatectomy

Exclusion Criteria:

* Chronic cardiac or pulmonary diseases

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of arterial oxygenation | at 6 hours (average duration of surgery procedure)

SECONDARY OUTCOMES:
evaluation of specific static elastance of the lung | at 6 hours (average duration of surgery procedure)
  Evaluation of the elastic properties of the lung (specific static elastance)
evaluation of difference between arterial end-tidal partial pressure of carbon dioxide | at 6 hours (average duration of surgery procedure)
  difference between arterial end-tidal partial pressure of carbon dioxide is an indicator of lung collapse and reopening after open-lung PEEP, which in turn reduce dead space

OTHER OUTCOMES:
variation of gas exchange in post operative period | at 1 week (average duration)

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Terragni, MD, Principal Investigator — University of Turin, Italy; Augusto Tempia, MD, Study Chair — University of Turin, Italy
Locations (1):
- A.O.U San Luigi Gonzaga Hospital, Univesity of Turin, Turin, Italy, Italy